CLINICAL TRIAL: NCT05509413
Title: DEFLAGYN® Vaginal Gel and Spontaneous Remission and Regression of Unclear Cervical Smears and HPV High-risk Infections
Acronym: HPV-VG1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Director, Department of Obstetrics and Gynecologiy, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPV-VG1
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cervix Dysplasia; HPV Infection
Keywords: cervical dysplasia; unclear cytology; HPV infection
MeSH Terms: conditions — Uterine Cervical Dysplasia; Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: 1:1 randomization into a control arm (wait-and-see) and a treatment arm (vaginal gel)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Wait-and-see approach.
- DEFLAGYN Arm (Experimental): Application of DEFLAGYN vaginal gel for 3x 28days (as per instructions provided by the manufacturer)
  Interventions: Device: DEFLAGYN vaginal gel

INTERVENTIONS:
Device: DEFLAGYN vaginal gel — DEFLAGYN is a vaginal gel, classified as a medical device, containing silica and citric acid, which binds pathogens, inhibits their spread and exerts an antioxidant effect. It is applied intravaginally (through an applicator) and used for 3 months.
  Arms: DEFLAGYN Arm

SUMMARY:
Human papillomaviruses (HPV) are the most common sexually transmitted pathogens worldwide and in most cases are causally associated with the development of cervical cancer, one of the most common cancers in women and one of the leading causes of death in women worldwide. Precancerous lesions (dysplasias) or the presence of a high-risk HPV subtype are detected by a screening smear test performed by a gynecologist. If precancerous lesions are detected, conization (= surgical removal of a cone of tissue from the cervix) is the method of choice for removing the diseased tissue. However, if the degree of dysplasia is correspondingly low or the smear is unclear, then the guideline-compliant non-surgical treatment provides for a wait-and-see approach with PAP and HPV smear control after 6-8 months.

This "wait-and-see" approach can be complemented by local therapy with an immunostimulant. For this purpose, DEFLAGYN® (a vaginal gel containing silica and citric acid) and Aldara® (imiquimod, a Toll-Like Re-ceptor 7 antagonist) are available. However, while the latter is not approved for the treatment of cervical dysplasia or HPV infection, DEFLAGYN® has CE marking and approval as a medical device for treatment in a number of indications, such as unclear cervical smears, HPV-induced cervical lesions, p16/Ki-67-positive cervical lesions or cervical erosions.

However, available studies on the efficacy of DEFLAGYN are limited. For example, there is only one prospective randomized trial (Major et al, 2021, Arch. Gynecol. Obstet. 303:501-511), which included 216 women with histologically confirmed CIN 1/2. A 3-month intravaginal application of DEFLAGYN® resulted in regression of CIN 1/2 in 72% versus 25% in the control arm (no intervention). Side effects of therapy with DEFLAGYN® were not observed in this study.

Due to the frequency of CIN and HPV infections in the female population and due to the high medical relevance of a conservative method of treating this disease, further methodologically high-quality studies on the efficacy of DEFLAGYN® should be performed.

DETAILED DESCRIPTION:
1. HPV and dysplasia of the cervix uteri Human papillomaviruses (HPV) are the most common sexually transmitted pathogens worldwide. The prevalence in both male and female populations is high. Epidemiological estimates suggest that 85-91% of sexually active adults acquire at least one genital HPV infection by age 50, with approximately 95% of HPV infections being spontaneously eliminated within 2 years in terms of HPV immunologic clearance. HPV preferentially infects the epithelial cells of the anogenital area and, through incorporation of HPV DNA into the host genome of the basal cells of the squamous epithelium of the cervix and subsequent expression of viral components, causes dysplastic changes in the cervical epithelium that, if left untreated, can develop into invasive carcinoma of the cervix (cervical carcinoma).

   Cervical carcinoma is the fourth most common cancer as well as the fourth leading cause of cancer-related death in women worldwide, responsible for 6.6% (570,000) of all new cancer cases and 7.5% (311,000) of cancer-related deaths in women in 2018.

   The precursor of squamous cell carcinoma of the uterine cervix (approximately 80% of all cervical cancers) is cervical intraepithelial neoplasia (CIN), which has three grades of expression (CIN1, CIN 2, and CIN 3). Compared with invasive cervical carcinoma, the incidence and prevalence of precancerous lesions of the cervix uteri are much higher. It is estimated that approximately 100,00 w0omen in Germany develop high-grade dysplasia (CIN2/CIN3) each year.
2. Therapy Dysplasia of the cervix typically becomes conspicuous during gynecological screening examinations. Here, smears are taken from the ectocervix and endocervix and assessed cytologically for dysplastic cells and the quality of the smear after Papanicolaou staining. HPV infection diagnostics are also performed as part of the statutory cervical carcinoma screening (annually or every 3 years) in order to detect the presence of HPV high risk infections.

   In case of abnormalities in the cervical smear and/or HPV high risk infection with suspicion of cervical dysplasia, presentation to a specialized dysplasia consultation is recommended for further clarification of dysplastic changes. During the subsequent colposcopic examination, a histological tissue sample ('cervical biopsy') of conspicuous areas is taken. The histopathological processing of the tissue samples and the colposcopic image of the spread of the changes in the cervix then allow individualized therapy planning.
3. Conization as the standard of surgical treatment If precancerous lesions with the potential to develop into an invasive cervical tumor are detected, conization (= surgical removal of a cone of tissue from the cervix) is the method of choice for removing the diseased tissue. The worldwide standard surgical procedure for conization is LLETZ conization (="Large Loop Excision of the Transformation Zone"). In addition to the risk of local persistence of precancerous lesions if cervical dysplasia is incompletely removed, LLETZ also increases the risk of preterm delivery in subsequent pregnancy. This risk increases with increasing volume of removed tissue. To reduce or avoid the aforementioned complications, conization should be performed under colposcopic vision and as little healthy cervical tissue as possible should be removed.
4. Non-surgical treatment options Non-surgical methods for the treatment of CIN and/or HPV high risk infections are limited. According to the current S3 guideline, in case of CIN 1 and/or HPV high risk infection, a wait-and-see approach with PAP and HPV smear control in 6-8 months is possible. Alternatively, local therapy with an immunostimulant may be used. DEFLAGYN® and Aldara® are available for this purpose. Aldara® is imiquimod, a Toll-Like Receptor 7 (TLR 7) antagonist, which leads to a local immune response. However, Aldara® is not approved for the treatment of CIN or HPV infections. DEFLAGYN®, on the other hand, has a CE mark and medical device approval for the treatment of unclear cervical smears (ASC-US, ASC-H, LSIL, HSIL or PAP II-p, PAP III-p, PAP IIID1, PAP IIID2 or PAP III, PAP IIID) or HPV-induced cervical lesions or p16/Ki-67-positive cervical lesions or cervical erosions.
5. DEFLAGYN® - Mode of action and approval status DEFLAGYN® is a vaginal gel containing silica and citric acid, which binds pathogens, inhibits their spread and exerts an antioxidant effect. It is applied intravaginally and used for 3 months. In a prospective randomized study of 216 women with histologically confirmed CIN 1/2, 3 months of intravaginal application of DEFLAGYN® resulted in regression of CIN 1/2 in 72% versus 25% in the control arm (no intervention). The rate of HPV high risk infections decreased from 87% to 44% in the intervention arm. No other intervention studies on the efficacy of DEFLAGYN® can be found in the literature (PubMed search on 08/14/2022; search terms: dysplasia, deflagyn, HPV, silicon dioxide gel, randomized). Side effects of therapy with DEFLAGYN® were not observed in the study. Due to the frequency of CIN and HPV infections in the female population and due to the high medical relevance of a conservative method of this disease, further methodologically high-quality studies on the efficacy of DEFLAGYN® are useful.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Unclear cervical smear (ASC-US, ASC-H, LSIL, HSIL or PAP II-p, PAP III-p, PAP IIID1, PAP IIID2 (Munich III) or PAP III, PAP IIID, PAP I + HPV high-risk infection)

Exclusion Criteria:

* Pregnancy
* Known hypersensitivity to any of the ingredients of the vaginal gel
* Insufficient knowledge of the German language
* Pre-existing oncological diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Rate of hr-HPV-positive cervical smears | 3 months after initial examination/study inclusion
  The rate of hr-HPV-positive findings after 3 months.

SECONDARY OUTCOMES:
Rate of hr-HPV-positive cervical smears | 6 months after initial examination/study inclusion
  The rate of hr-HPV-positive findings after 6 months.
Rate of progression | 3 and 6 months after initial examination/study inclusion
  The rate of progression (in case of mild dysplasia at start)
Rate of newly diagnosed dysplasia | 3 and 6 months after initial examination/study inclusion
  The rates of newly diagnosed (i.e. not present during initial examination at study start) dysplasia or malignancies
Complications | From study inclusion/treatment start until the 3-month-follow up visit
  The number and kind of complications during the first 3 months

OTHER OUTCOMES:
Patients' Satisfaction | 3 and 6 months after initial examination/study inclusion
  General satisfaction of the patients with quality of care (100-mm-visual analog scale; 0 = very unsatisfied, 100=very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Clemens B Tempfer, MD, MBA, Principal Investigator — Ruhr-Universität Bochum, Marien Hospital Herne
Locations (1):
- Marien Hospital Herne, Herne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request made to the corresponding author. This includes individual participant data underlying the results presented here, after deidentification, as well as data dictionaries and the the study protocol. Data is available after publication, without a specific end date. Requesting investigators must show that their proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication of the study results, no time limit.
Access Criteria: Reasonable request, approval of the intended study by an independent review committee identified for this purpose.

REFERENCES:
- [Background] Workowski KA, Bachmann LH, Chan PA, Johnston CM, Muzny CA, Park I, Reno H, Zenilman JM, Bolan GA. Sexually Transmitted Infections Treatment Guidelines, 2021. MMWR Recomm Rep. 2021 Jul 23;70(4):1-187. doi: 10.15585/mmwr.rr7004a1. PMID 34292926
- [Background] Chesson HW, Dunne EF, Hariri S, Markowitz LE. The estimated lifetime probability of acquiring human papillomavirus in the United States. Sex Transm Dis. 2014 Nov;41(11):660-4. doi: 10.1097/OLQ.0000000000000193. PMID 25299412
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Mathevet P, Chemali E, Roy M, Dargent D. Long-term outcome of a randomized study comparing three techniques of conization: cold knife, laser, and LEEP. Eur J Obstet Gynecol Reprod Biol. 2003 Feb 10;106(2):214-8. doi: 10.1016/s0301-2115(02)00245-2. PMID 12551795
- [Background] Bevis KS, Biggio JR. Cervical conization and the risk of preterm delivery. Am J Obstet Gynecol. 2011 Jul;205(1):19-27. doi: 10.1016/j.ajog.2011.01.003. Epub 2011 Feb 23. PMID 21345402
- [Background] Jin G, LanLan Z, Li C, Dan Z. Pregnancy outcome following loop electrosurgical excision procedure (LEEP) a systematic review and meta-analysis. Arch Gynecol Obstet. 2014 Jan;289(1):85-99. doi: 10.1007/s00404-013-2955-0. Epub 2013 Jul 11. PMID 23843155
- [Background] Khalid S, Dimitriou E, Conroy R, Paraskevaidis E, Kyrgiou M, Harrity C, Arbyn M, Prendiville W. The thickness and volume of LLETZ specimens can predict the relative risk of pregnancy-related morbidity. BJOG. 2012 May;119(6):685-91. doi: 10.1111/j.1471-0528.2011.03252.x. Epub 2012 Feb 14. PMID 22329499
- [Background] Shaco-Levy R, Eger G, Dreiher J, Benharroch D, Meirovitz M. Positive margin status in uterine cervix cone specimens is associated with persistent/recurrent high-grade dysplasia. Int J Gynecol Pathol. 2014 Jan;33(1):83-8. doi: 10.1097/PGP.0b013e3182763158. PMID 24300540
- [Background] Preaubert L, Gondry J, Mancini J, Chevreau J, Lamblin G, Atallah A, Lavoue V, Caradec C, Baldauf JJ, Bryand A, Henno S, Villeret J, Agostini A, Douvier S, Jarniat A, Riethmuller D, Mendel A, Brun JL, Rakotomahenina H, Carcopino X. Benefits of Direct Colposcopic Vision for Optimal LLETZ Procedure: A Prospective Multicenter Study. J Low Genit Tract Dis. 2016 Jan;20(1):15-21. doi: 10.1097/LGT.0000000000000156. PMID 26704328
- [Background] Kuhn W. [Colposcopy in the diagnosis of early cervical cancer]. Pathologe. 2011 Nov;32(6):497-504. doi: 10.1007/s00292-011-1480-9. German. PMID 21984389
- [Background] Major AL, Dvorak V, Schwarzova J, Skrivanek A, Malik T, Pluta M, Mayboroda I, Grandjean EM. Efficacy and safety of an adsorbent and anti-oxidative vaginal gel on CIN1 and 2, on high-risk HPV, and on p16/Ki-67: a randomized controlled trial. Arch Gynecol Obstet. 2021 Feb;303(2):501-511. doi: 10.1007/s00404-020-05816-8. Epub 2020 Nov 20. PMID 33219482
- [Background] Major AL, Skrivanek A, Grandjean EM, Dvorak V, Malik T, Pluta M, Mayboroda I. An Adsorptive and Antioxidant Vaginal Gel Clears High-Risk HPV- and p16/Ki-67-Associated Abnormal Cytological Cervical Findings: A post-hoc Subgroup Analysis of a Prospective Randomized Controlled Trial on CIN2 and p16 Positive CIN1. Front Med (Lausanne). 2021 May 25;8:645559. doi: 10.3389/fmed.2021.645559. eCollection 2021. PMID 34113633
- See also: German S3 Guidelines — https://www.leitlinienprogramm-onkologie.de/leitlinien/zervixkarzinom-praevention/